CLINICAL TRIAL: NCT01989845
Title: Prospective, Multicenter Study Investigating Efficacy and Safety of Oral Rivaroxaban for the Prevention of Recurrent Venous Thromboembolism in Korean Patients With Cancers
Brief Title: Rivaroxaban for the Prevention of Venous Thromboembolism in Asian Patients With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Society of Hematology Thrombosis Working Party (Unknown)
Responsible Party: Principal Investigator, Soo-Mee Bang, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KVTE13-01
Record Dates: First submitted 2013-11-05; First posted 2013-11-21 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Rivaroxaban; Cancer-associated Thrombosis; Recurrence; Bleeding
MeSH Terms: conditions — Recurrence; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral rivaroxaban in cancer-associated VTE (Experimental)
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15mg twice daily for the first 3 weeks, followed by 20mg once daily during 6 months
  Other Names: Xarelto

SUMMARY:
Rivaroxaban has been developed in the various clinical settings, prevention of venous thromboembolism (VTE)after major orthopedic surgery, prevention of stroke in atrial fibrillation, and in the treatment of acute coronary syndromes. And, in the EINSTEIN-pulmonary embolism (PE) and EINSTEIN-deep venous thrombosis (DVT) programs, rivaroxaban showed non-inferior to standard therapy for the treatment of PE and DVT. However, there has been limited experience of rivaroxaban with secondary VTE prophylaxis in cancer patients. Although cancer-associated DVT or PE was included in previously mentioned EINSTEIN programs, only approximately 5% of the total populations were cancer patients in these studies. Thus, investigators could not automatically translate the results of these studies into the real practice management of cancer-associated VTE patients. Moreover, until now, new oral anticoagulants, including dabigatran and rivaroxaban, have been compared to long-term warfarin therapy, which were well-known inferior agent, but not low molecular weight heparin. In this sense, investigators feel that new oral anticoagulants, particularly rivaroxaban, should be re-investigated in this highly specific patients group. Therefore, investigators are planning to conduct a prospective study evaluating the efficacy and safety of rivaroxaban in Korean patients with cancer-associated VTE.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old and active cancer and newly-diagnosed, symptomatic or incidental proximal lower extremity DVT, PE or both
* will have a life expectancy > 3 months
* will be treated with anticoagulation therapy for at least 3 months.

Exclusion Criteria:

* (1) Isolated asymptomatic distal DVT
* (2) Intra-abdominal venous thrombosis or vascular access-induced thrombosis
* (3) Hemodynamically unstable PE, indicating systolic blood pressure <90 mmHg
* (4)Eastern Cooperative Oncology Group (ECOG) performance status score of 3 or 4
* (5) History of total gastrectomy
* (6) Overt brain metastasis. Patients who have controlled brain metastasis without need of glucocorticoid are eligible
* (7) History of recent major or clinically relevant bleeding within the previous 4 weeks
* (8) Conditions associated with a high risk of serious bleeding (active peptic ulcer or recent neurosurgery)
* (9) Other serious illness or medical conditions (illnesses requiring chronic anticoagulation therapy, unstable cardiac disease despite treatment, myocardial infarction within 3 months prior to study entry, significant neurologic or psychiatric diseases including dementia or seizure, active uncontrolled infection, other serious medical conditions)
* (10)Inadequate renal function; creatinine clearance < 30 ml/min
* (11) Inadequate hepatic function: alanine aminotransferase > 3 times the upper limit of normal (ULN) (if liver metastasis, alanine aminotransferase > 5 times the ULN or total bilirubin >2 times the ULN (if liver metastasis, total bilirubin >3 times the ULN)
* (12) Baseline platelet count < 75,000 per cubic millimeter or Hb < 8g/dL
* (13) Plan of treatment with bevacizumab or other anti-cancer drugs known to increase the bleeding risk
* (14) Women of childbearing potential who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period, who are using a prohibited contraceptive method, or who are pregnant or breastfeeding
* (15) Patients requiring strong cytochrome P450 3A4 (CYP3A4) inducers (rifampin, phenobarbital) or strong CYP3A4 inhibitors (HIV protease inhibitor, systemic ketoconazole) treatments
* (16) Patients with inferior vena cava filter placement or underwent catheter-directed thrombolysis or stent placement for the treatment of index VTE

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
recurrent symptomatic deep venous thrombosis, pulmonary embolism or both | within the six months after the diagnosis of index VTE
  Recurrent DVT will be defined if a new onset non-compressibility of a previously compressible venous segment on ultrasonography is identified or if there is a new constant intraluminal filling defect on venography. Unequivocal extension of the thrombus will be needed to diagnose the recurrence on the same extremity of the first event unless new concomitant PE or DVT in other extremities is confirmed.
  Recurrent PE will be diagnosed by high probability on ventilation/perfusion lung scan, or by the presence of non-enhancing filling defects in the pulmonary vasculature on pulmonary CT angiogram.

SECONDARY OUTCOMES:
incidentally detected VTE | within six months after the diagnosis of VTE
  Incidentally detected recurrent thrombosis will be defined as objectively-proven thrombosis during the study period by imaging studies that are performed for reasons other than suspected VTE.
Major or clinically relevant non-major bleedings | within six months after the diagnosis of VTE
  Major bleeding will be defined if it is associated with death, occurs at critical sites (intracranial, intraspinal, intraocular, retroperitoneal, or pericardial area), and results in a need for a transfusion of at least 2 units of packed red cells, or lead to a drop in hemoglobin of more than 2 g/dL.
  Clinically relevant non-major bleeding will be defined as relevant bleeding that did not meet the criteria for major bleeding but is associated with medical intervention, unscheduled visit, interruption or discontinuation of a study drug, or discomfort or impairment of activities of daily life
recurrent VTE according to the risk of clinical prediction rule | within six months after the diagnosis of VTE
  Risk of recurrent VTE can be differentiated by risk prediction rule, named Ottawa score. Ottawa score is composed of gender, primary tumor site, stage, and prior VTE and ranged between -3 and 3 score points. Patients with a score <1 will be considered as having low risk for recurrence and patients with a score >1 considered as having high risk for recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Mee Bang, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea